CLINICAL TRIAL: NCT03519620
Title: The Effects of Swimming and Swimming Complemented With Water Walking on Spirometry Values
Brief Title: Swimming and Water Walking on Spirometry Values
Acronym: ESWWSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Collaborators: Municipal Swimming Clube (Unknown)
Responsible Party: Principal Investigator, Samuel Honório, Principal Investigator, Instituto Politécnico de Castelo Branco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPCB
Record Dates: First submitted 2018-04-16; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Child Development; Child Obesity; BMI
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SWWSV (Experimental): Spirometric Values: Forced Vital Capacity; Forced Expiratory Volume in 1 second; Peak Expiratory Flow
  Interventions: Other: SWWSV

INTERVENTIONS:
Other: SWWSV — Behaviours to prevent child obesity

SUMMARY:
To study the effects of swimming with water walking in children aged between 6 and 12 years in terms of spirometric values.

DETAILED DESCRIPTION:
The present research aims to verify if there are differences in body composition and spirometric values in children aged between 6 and 12 years who practice swimming complemented with water walking at the end of each session and those who only practice swimming. The sample consisted of 28 individuals aged 6 to 12 years and was divided into two groups: swimming group (SG) with 9 children and swimming complemented with water walking group (SWWG) of 19 children. In this study, the investigators wanted to know which were the benefits in body composition and for that purpose used a bio-impedance scale Targa Silvercrest Z29777A (Germany), and an anthropometric tape to measure the waist circumference. To calculate the spirometric values, namely forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and even peak expiratory flow (PEF) a Cosmed Microquark spirometer was used. In terms of statistical procedures, the investigators used the program Statistical Package for the Social Sciences version number 20 (SPSS 20.0). The investigators used descriptive statistics (minimum, maximum, means and standard deviations), the Shapiro Wilk test for testing the normality of the sample, inferential statistics (non-parametric Mann-Whitney tests, Friedman's Anova, and for the calculation of the effect magnitude the d-Cohen test). After the data treatment, regarding the inter-group analysis (comparison between the swimming group and the swimming group with water walking) the investigators observed that there were significant differences in three variables at the end of the study, that is, at the end of the 3 moments. These variables were weight relative to body composition, forced expiratory volume in 1 second (FEV1) and peak expiratory flow (PEF), these values are relative to the spirometry evaluation. Concerning intra-group differences (improvement in the swimming group and the swimming with water walking group in the three moments evaluated), the SWWG showed significant improvements in the variables of weight, muscle mass, fat mass, percentage of water, body mass index (BMI), body percentiles, forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* Children inside this age range;
* water experience between 6 and 12 months
* children with no other activities besides swimming

Exclusion Criteria:

* Children with Asma;
* Children with DPOC
* Children with pulmonary limitations.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity | 12 weeks
  described in liters
Forced Expiratory Volume in 1 second | 12 weeks
  described in liters
Peak Expiratory Flow | 12 weeks
  described in liters

SECONDARY OUTCOMES:
Fat mass | 12 weeks
  described in percentage
Weight | 12 weeks
  described in kilograms
Height | 12 weeks
  described in meters
weight and height will be combined to report BMI | 12 weeks
  BMI described in kg/m^2
Muscle mass | 12 weeks
  described in percentage
waist circumference | 12 weeks
  described in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: João B Oliveira, Master, Principal Investigator — Castelo BRanco
Locations (1):
- Municipal Swimming Pools, Castelo Branco, Portugal

IPD SHARING:
Plan to Share IPD: No